CLINICAL TRIAL: NCT02878798
Title: Topiramate as a Disease Modifying Therapy for Cryptogenic Sensory Peripheral Neuropathy in Metabolic Syndrome (CSPN)
Brief Title: Topiramate for Cryptogenic Sensory Peripheral Neuropathy in Metabolic Syndrome (CSPN)
Acronym: TopCSPN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); NeuroNEXT Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URNN001 / HM20014083; 1U01NS095388 (NIH)
Record Dates: First submitted 2016-08-11; First posted 2016-08-25 (Estimated); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Cryptogenic Sensory Peripheral Neuropathy in Metabolic Syndrome
MeSH Terms: interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): An overencapsulated placebo of identical color, shape and packaging to topiramate will be used.
  Interventions: Other: Placebo
- Topiramate (Experimental): Oral topiramate
  Interventions: Drug: topiramate

INTERVENTIONS:
Drug: topiramate — Oral topiramate at a target dose of 50mg twice daily.
  Other Names: Topamax
  Arms: Topiramate
Other: Placebo — overencapsulated placebo of identical color, shape and packaging to topiramate
  Arms: Placebo

SUMMARY:
The TopCSPN trial is a double blinded randomized placebo controlled study of oral topiramate as a potential disease modifying therapy for cryptogenic sensory peripheral neuropathy (CSPN). Patients with CSPN who also have metabolic syndrome (defined by the ATPIII criteria) who do not have an alternative cause for neuropathy will be potentially eligible. The co primary outcome measures are change in the Norfolk Quality of Life - Diabetic Neuropathy (NQOL-DN) Scale and intraepidermal nerve fiber density (IEFND) at the distal thigh. The treatment phase will last 24 months.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-80
2. Diagnosis of confirmed symptomatic distal symmetric peripheral polyneuropathy based on the Toronto consensus criteria for probable neuropathy (the presence of unequivocal signs and symptoms of neuropathy)45.
3. Evidence of symptomatic neuropathy based on a screening visit NQOL-DN score of >9.
4. Metabolic syndrome based on modified ATPIII criteria. Specific criteria require 3 of the following 6 to be present at the screening visit.

   * Waist circumference >102 cm for men, >88 cm for women
   * Serum triglycerides of > 150 mg/dl
   * HDL < 40 mg/dl for men, < 50 mg/dl for women
   * Those with either a normal HDL or TRG who are taking a lipid lowering medication for this purpose
   * Blood pressure 130/85 mm Hg or use of anti-hypertension drug
   * Hyperglycemia based on American Diabetes Association (ADA) criteria at screening based on any one or more of the following: fasting plasma glucose > 100 mg/dL (5.6 mmol/L), 2-hour glucose tolerance test > 140 mg/dL (7.8 mmol/L), or hemoglobin A1c > 5.7% .
5. No current or prior history of therapy with topiramate.
6. If female of child-bearing potential (i.e., not surgically sterile or post-menopausal defined as age > 51 years without menses for ≥ 2 years), negative serum pregnancy test at screening and negative urine pregnancy test at baseline visit.
7. Women of child-bearing potential or men with sexual partners of childbearing potential be willing to use an acceptable method of birth control for the duration of the study and for 12 weeks following completion of study drug therapy. Acceptable methods of birth control include abstinence, oral contraceptives, the contraceptive patch, intra-uterine device, the contraceptive ring, and or barrier contraception such as condoms with spermicide.

Exclusion Criteria

1. CSS-PI clinical determination of an alternative cause for peripheral neuropathy (including but not limited to rheumatological disorders, Hepatitis B or C, breast cancer treated with neurotoxic chemotherapy within the past 15 years). All potential subjects will have screening neuropathy labs including assessment for diabetes (Hemoglobin A1c, oral glucose tolerance test), vitamin B12 level, and immunofixation47.
2. Type I diabetes or current use of insulin or use of insulin in the past 3 months.
3. HgA1c > 7.5%. Borderline screening labs can be repeated within two weeks with PPI approval.
4. History of recurrent nephrolithiasis, a single episode of nephrolithiasis within one year prior to screening, or use of ongoing preventative treatment.
5. Family history of a hereditary neuropathy in a first-degree relative.
6. Severe neuropathy: Utah Early Neuropathy Score > 24 at screening
7. Active foot ulceration or a history of a nontraumatic foot amputation.
8. ECG with QTc more than 450 ms in men, or 470 ms in women.
9. Risk of excessive bleeding at the skin biopsy site based on the clinical assessment of the CSS-PI.
10. Chronic corticosteroid use excluding topical or inhaled treatment.
11. Use of a carbonic anhydrase inhibitor (such as acetazolamide) due to risk of nephrolithiasis.
12. Planned bariatric surgery.
13. Use of other weight loss medications.
14. Use of scheduled opiates, or as needed opiate medications more than three times weekly.
15. Use of topical capsaicin products within 16 weeks of screening or at any time on study.
16. Medication change for neuropathy symptoms during the 8 weeks prior to screening; or anticipated change for the duration of study participation.
17. Current use of an intrathecal pain pump or spinal cord stimulator.
18. Screening laboratory creatinine ≥ 2.0 mg/dl.
19. Severe edema, dermatologic or lower extremity condition that would increase risk of skin biopsy.
20. Major depression, bipolar affective disorder, or other mental health disorders that are sufficiently severe to increase adverse event risk or impact neuropathy assessment in the opinion of the responsible site principal investigator.
21. Current suicidal ideation within one year prior to the baseline visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS).
22. Ataxia sufficiently severe to represent an unacceptable fall risk in the opinion of the site principal investigator.
23. A serious medical condition expected to dramatically shorten life span or prevent participation.
24. Any clinically significant condition or illness, which, in the opinion of the CSS-PI, would pose a risk to the subject or might confound the study including metabolic acidosis, bone marrow suppression, blood dyscrasias, bleeding disorder, or closed angle glaucoma.
25. History of alcohol or drug abuse within the past two years, or existing neuropathy related to past drug or alcohol abuse.
26. History of malignancy within five years prior to study enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
27. A history of epilepsy.
28. An inability to understand or cooperate with the procedures of the study.
29. Pregnant, or intending to become pregnant, or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Smith, MD, Principal Investigator — Virginia Commonwealth University
Locations (20):
- United States (20):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Neurology Clinical Trials Organization, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical Center, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith AG, Singleton JR, Aperghis A, Coffey CS, Creigh P, Cudkowicz M, Conwit R, Ecklund D, Fedler JK, Gudjonsdottir A, Hauer P, Herrmann DN, Kearney M, Kissel J, Klingner E, Quick A, Revere C, Stino A; NeuroNEXT NN108 TopCSPN Study Team. Safety and Efficacy of Topiramate in Individuals With Cryptogenic Sensory Peripheral Neuropathy With Metabolic Syndrome: The TopCSPN Randomized Clinical Trial. JAMA Neurol. 2023 Dec 1;80(12):1334-1343. doi: 10.1001/jamaneurol.2023.3711. PMID 37870862

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Topiramate
Started | 66 | 66
Completed | 59 | 59
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Topiramate | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.7) | 61.9 (9.9) | 62.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 44 | 38 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 62 | 66 | 128
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 60 | 62 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Intraepidermal Nerve Fiber Density (IENFD)
Description: Difference in IENFD change between treatment groups over 96 weeks (fibers/mm) (i.e. the slope of change). A skin biopsy is obtained. The sample is stained for nerve fibers. The rate of change in IENFD in fibers/mm is calculated over the 96 week duration of the study and expressed in change in fibers/mm/year (defined as 52 weeks) over the study period (i.e. the slope of change expressed and change in IENFD in fibers/mm over a 52 week period).
Time Frame: 96 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: fibers/mm/year (52 weeks)
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
fibers/mm/year (52 weeks) | -0.6064 [-1.1785 to -0.03437] | -0.396 [-0.9625 to 0.1705]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Other — Non-inferiority and superiority tests were completed; Slope = 0.2105, 95% CI 1-sided [lower limit -0.4328]

2. Primary Outcome: Norfolk Quality of Life - Diabetic Neuropathy
Description: Difference in NQOL between treatment groups over 96 weeks. The Norfolk QOL-DN is a validated 47-item, patient-reported outcome measure, sensitive to the different features of diabetic neuropathy (DN) including small fiber, large fiber, and autonomic function. A lower score is better. The range of the score is from -4 to 136. The slope of the change in total Norfolk QOL-DD is calculated as the change in total score/52 weeks (one year)
Time Frame: 96 weeks (expressed as a slope in change of total score/52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Change inTotal NQOL-DN score over 52 wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
Change inTotal NQOL-DN score over 52 wks | 3.5815 [1.3162 to 5.8467] | 2.0596 [-0.2545 to 4.3737]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Other — Non-inferiority and superiority tests were done; Slope = -1.5219, 95% CI 1-sided [upper limit 1.1933]

3. Secondary Outcome: Brief Pain Inventory - Diabetic Neuropathy (BPI-DN) Pain Interference
Description: Pain interference score. Each item is scored from 0-10 with a total possible number of points of 70, higher worse. The range of the score is 0-70. The change in score is expressed as a slope of change in pain interference score/52 weeks (one year)
Time Frame: 96 weeks (expressed as a change in change in pain interference/52weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Slope of change in BPI-DN PI over 52 wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
Slope of change in BPI-DN PI over 52 wks | 0.1999 [-0.3602 to 0.7600] | 0.1767 [-0.3984 to 0.7517]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; Mixed Models Analysis; Slope = -0.02322, 95% CI 2-sided [-0.6337 to 0.5872]

4. Secondary Outcome: Brief Pain Inventory - Diabetic Neuropathy (BPI-DN) Average Pain Intensity
Description: Average pain severity. Each item is scored 0-10 with a total of 40 possible points, higher is worse. The range of the score is 0-40. The slope of the change in this score is expressed as change/one year (defined as 52 weeks)
Time Frame: 96 weeks (expressed as a slope of change over 52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Slope of change in BPI-DN pain over 52 w
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
Slope of change in BPI-DN pain over 52 w | -0.1046 [-0.3431 to 0.1338] | -0.2726 [-0.5176 to -0.0276]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.261, Mixed Models Analysis; Slope = -0.168, 95% CI 2-sided [-0.4612 to 0.1253]

5. Secondary Outcome: Utah Early Neuropathy Scale
Description: The UENS is a validated examination score of neuropathy severity based on a physical examination (Singleton et al 2008). Total score is 42 (minimum 0 and maximum 42). The higher the score, the worse the outcome is. The change in UENS over the 96 week period is expressed as a slope of change in total UENS over one year defined as 52 weeks.
Time Frame: 96 weeks (expressed as a slope of change in total UENS over 52 weeks).
Measure: Least Squares Mean (95% Confidence Interval); unit: Slope of change in Total UENS over 52wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
Slope of change in Total UENS over 52wks | 0.4281 [-0.2409 to 1.0970] | 0.3671 [-0.3220 to 1.0562]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.9007, Mixed Models Analysis; Slope = -0.061, 95% CI 2-sided [-1.0213 to 0.8992]

6. Secondary Outcome: Sural Sensory Amplitude (SSA)
Description: Change in SSA measured in microvolts. SSA is measured by electrically stimulating a nerve through the skin and recording the response. A larger value is better. The normal values vary based on age, with a minimum of 0 (absent). Across all ages, the lower limit of normal is 6 microvolts, although the normal cutoff declines with aging. The change in SSA over the 96 week study period is expressed as a slope of change in uV/52 weeks (the 52 week log (mV) change of non-zero values).
Time Frame: 96 weeks (slope of change in mV/52weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: slope of change in SSA uV over 52 wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
slope of change in SSA uV over 52 wks | 0.0334 [-0.0320 to 0.0987] | 0.044 [-0.0232 to 0.1111]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.8174, Hurdle model; Slope = 0.0106, 95% CI 2-sided [-0.0793 to 0.1005]

7. Secondary Outcome: Peroneal Motor Conduction Velocity (PMCV)
Description: PMCV change. PMCV is measured by electrically stimulating the nerve through the skin at two different locations and measuring how fast the response travels between the two in meters/second. A higher value is better. The slope of the change in PMCV is expressed as change in meters/second/52 weeks (one year).
Time Frame: 96 weeks (expressed as a slope of change in meter/sec over 52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Slope of change in M/S over 52 wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 60 | 63
Slope of change in M/S over 52 wks | -0.04363 [-0.5073 to 0.4200] | -0.783 [-1.2347 to -0.3314]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.0233, Mixed Models Analysis; Slope = -0.7394, 95% CI 2-sided [-1.3775 to -0.1013]

8. Secondary Outcome: Body Mass Index (BMI)
Description: BMI change in kg/m2. BMI is a measure of weight relative to height. The slope of the change in BMI over the study was expressed as change in kg/m2/52 weeks.
Time Frame: 96 weeks (slope of change in kg/m2/52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Slope of change in BMI kg/m2 over 52wks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
Slope of change in BMI kg/m2 over 52wks | -0.1537 [-0.7461 to 0.4387] | -0.2865 [-0.8952 to 0.3221]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.7586, Mixed Models Analysis; Slope = -0.1328, 95% CI 2-sided [-0.982 to 0.7164]

9. Secondary Outcome: Hemoglobin A1C
Description: Slope of the Hemoglobin A1C change. A1C is measured in percent. It provides an estimate of how high blood sugar has been over the past three months. A higher value indicates poor diabetic control.
Time Frame: The annual slope of the change in A1C over 96 weeks expressed in change in percent/52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: change in %/52 weeks over 96 weeks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
change in %/52 weeks over 96 weeks | 0.03 [-0.0281 to 0.0880] | 0.0279 [-0.0299 to 0.0858]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.9604, Mixed Models Analysis; Slope = -0.0021, 95% CI 2-sided [-0.084 to 0.0799]

10. Secondary Outcome: Serum Triglycerides (TRG)
Description: TRG change. TRG are a type of lipid or fat circulating in the blood. A higher value is associated with increased cardiovascular risk. The slope of the change in TRG was calculated as change in mg/dl over 52 weeks (one year).
Time Frame: 96 weeks (slope of change mg/dl over 52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: change in mg/dl/52 weeks over 96 weeks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
change in mg/dl/52 weeks over 96 weeks | 0.022 [-0.0258 to 0.0698] | -0.0176 [-0.0654 to 0.0301]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.2365, Mixed Models Analysis; Slope = -0.0396, 95% CI 2-sided [-0.1053 to 0.0261]

11. Secondary Outcome: LDL Cholesterol
Description: LDL change. LDL is "bad" cholesterol, measured in mg/dL. A higher value is associated with elevated cardiovascular risk. A slope of change is calculated change in LDL in mg/dL/52 weeks (one year)
Time Frame: 96 weeks (expressed as a slope of change in mg/dl/52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: change in mg/dl/52 weeks at 96 weeks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
change in mg/dl/52 weeks at 96 weeks | -6.6584 [-12.7056 to -0.6112] | -4.2736 [-10.3001 to 1.7529]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.5813, Mixed Models Analysis; Slope = 2.3848, 95% CI 2-sided [-6.1336 to 10.9032]

12. Secondary Outcome: HDL Cholesterol
Description: HDL change. HDL is "good cholesterol", measured in mg/dL. A lower value is associated with higher cardiovascular risk. The slope of change is calculated as change in mg/dL/52 weeks (one year)
Time Frame: 96 weeks (expressed as slope of change in mg/dL/52 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: change in mg/dl/52 weeks at 96 weeks
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 66 | 66
change in mg/dl/52 weeks at 96 weeks | 0.8156 [-0.9673 to 2.5985] | -0.2391 [-2.0143 to 1.5361]
Statistical Analysis 1: Comparison: Placebo vs Topiramate; Test type: Superiority; p = 0.4092, Mixed Models Analysis; Slope = -1.0547, 95% CI 2-sided [-3.5705 to 1.4611]

ADVERSE EVENTS:
Time Frame: Participants will be monitored for AEs from the time they sign consent until 30 days following permanent discontinuation of study drug.
Description: If an observed or reported sign, symptom, or clinically significant (CS) laboratory anomaly is not considered by the Site Investigator to be a component of a specific disease or syndrome, then it should be recorded as a separate AE on the AE CRF. CS laboratory abnormalities, such as those that require intervention, are those that are identified as such by the Site Investigator.
Arm/Group | Placebo | Topiramate
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 9/66 | 4/66
Other Adverse Events (participants affected / at risk) | 56/66 | 61/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Topiramate (N=66)
Cataract (Eye disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Aortic Aneurysm (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Decubitis Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dressler's Syndrome (Cardiac disorders) | 1 | 0
Lumbar Spinal Stenosis (Nervous system disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Non-Small Cell Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Parathyroidectomy (Surgical and medical procedures) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Localized Infection (Infections and infestations) | 0 | 1
Osteotomy (Surgical and medical procedures) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Topiramate (N=66)
Diarrhea (Gastrointestinal disorders) | 7 | 10
Dry Mouth (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 2 | 6
Fatigue (General disorders) | 5 | 13
Sinusitis (Infections and infestations) | 4 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Cognitive Disorder (Nervous system disorders) | 0 | 9
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 4 | 5
Memory Impairment (Nervous system disorders) | 1 | 6
Neuropathy Peripheral (Nervous system disorders) | 5 | 4
Paraesthesia (Nervous system disorders) | 9 | 14
Tremor (Nervous system disorders) | 3 | 4
Anxiety (Psychiatric disorders) | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7
Dysgeusia (Nervous system disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02878798/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT02878798/ICF_000.pdf